CLINICAL TRIAL: NCT01605188
Title: Predictors of Non-response and Loss of Response in IBD Patients Treated With Anti-TNF.
Status: Completed | Type: Observational
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Nikos Viazis, Consaltant Gastroenterologist, Evangelismos Hospital
Other Study IDs: nviazis2
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Serum Bowel mucosal tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of our study is to prospectively identify, at diagnosis, factors predictive of non-response or loss of response in patients with inflammatory bowel disease treated with anti-TNF.

DETAILED DESCRIPTION:
Crohn's disease and ulcerative colitis are both chronic idiopathic inflammatory conditions of the gastrointestinal tract that result in a considerably decreased quality of life. Long term experience with standard therapies for inflammatory bowel disease patients up to the late 1990s demonstrated diverse limitations. Corticosteroids have good short term efficacy, but are not suitable for maintaining remission, while treatment with immunomodulators are associated with an important risk of side effects. The introduction of monoclonal antibody to tumor necrosis factor a (TNFa) therapy has offered new treatment options originally in patients with Crohn's disease and more recently in those with ulcerative colitis as well. Several clinicians based on the results of clinical trials, now advocate the early use of intensive therapy (immunosuppressants and/or biologics) to maintain a good quality of life from the first flare up and prevent any irreversible consequence of the disease.

In 1998 infliximab was the first anti-TNF therapy to be approved by the U.S. Food and Drug Administration (FDA) for the treatment of adult patients with moderately to severely active luminal and fistulizing CD who have an inadequate response to conventional therapies. In 2007 adalimumab was also approved for the treatment of adult patients with moderate to severe CD. More recently, infliximab has been approved for the treatment of ulcerative colitis patients. The current recommendation for infliximab dosing comprises induction with 5 mg/kg at 0, 2, and 6 weeks, followed by maintenance 5 mg/kg every 8 weeks. Adalimumab is administered at a dose of 160 mg initially followed by 80 mg 2 weeks later and then at a dose of 40 mg every other week.

Since the aim of administering anti-TNF therapy is achieving disease remission, it should be noted that in the clinical setting, remission is defined as the absence of any gut-related symptoms, with a normal C-reactive protein (CRP) or erythrocyte sedimentation ratio (ESR), hemoglobin, albumin, and platelet count. Clinical response is defined as the improvement of symptoms (reduced bowel frequency, reduced urgency, improved stool consistency, reduced abdominal pain, reduced rectal bleeding, improved general well-being, increased energy, and reduced lethargy) and improvement in blood test parameters (reduced CRP, ESR, and platelet count, and improved albumin and hemoglobin).

Despite the high response rate, some patients do not improve after initiation of anti-TNF therapy or worsen after initial response. In the ACCENT I trial, 42% of patients had a primary lack of response to infliximab induction therapy, while in the CHARM trial, 42% of patients had a primary non-response to open label adalimumab induction therapy. According to literature data, diminished or complete loss of initial response to anti-TNF therapy can occur at any time after treatment begins and can occur at 30-50% of the patients treated. Regaining response can be achieved by either reducing the frequency of infusions or by increasing the dose, whether sometimes an increase of the dose plus a reduction of the dose interval is required.

Primary non-response is defined as the lack of response or minimal, clinically insignificant response after initiation of a biological agent. To be defined as demonstrating primary non-response a patient should have objective evidence of active inflammation and symptoms related to IBD. There is currently no consensus on how long a biological drug should be continued before lack of response is declared, although 58% of patients who will demonstrate a response to infliximab do so within 2 weeks. A substantial proportion of patients, however, will demonstrate a response up to 12 weeks after commencing treatment. Most responders demonstrate a clinical response by week 14 (in the case of infliximab that usually includes three induction plus one further dose). With adalimumab induction therapy it may require up to 12 weeks to determine whether response has been achieved. Loss of response is defined as an initial response to a biological drug followed by a diminished or less durable response over time.

For CD patients, primary non-response has been defined variously as failure to achieve a defined fall of CDAI from baseline, or a CDAI which remains greater than 220. Loss of response has been defined by a CDAI of greater than 220, which correlates with at least mild disease activity. In patients with primary non-response, or loss of response, to an anti-TNF drug, consideration should be given to reassessing disease activity and excluding complications such as the development of stenosing disease, an abscess, or infections, including cytomegalovirus and Clostridium difficile.

Given the morbidity associated with inappropriate dosing and the high costs associated with therapy with biologic agents, determining predictors of non-response of loss of response (need for dose escalation) has important clinical and economic implications. However, there exists a paucity of research examining such factors.

Endoscopy (ileocolonoscopy) will be performed at baseline (i.e. before anti-TNF administration) for all patients included in the study. For Crohn's disease patients, the simplified endoscopic severity index will be recorded (SES-CD), table 1, while the CD activity index (CDAI) will also be determined. For ulcerative colitis, the Mayo endoscopic subscore will be recorded (0: normal mucosa, 1: faded vascular pattern, mild friability, 2: loss of vascular pattern, erosions, friability, 3: ulcers of spontaneous bleeding). Disease activity will be graded according to the Clinical Activity Index (Lichtiger's CAI), with a highest possible score of 21. For all ulcerative colitis patients the Montreal classification of the extent of the disease will also be assessed.

Laboratory data on blood hemoglobin, hematocrit, white blood cells, plasma or serum albumin and C-reactive protein will be collected for all patients at baseline. Use of concurrent medication will be recorded, especially the dosage data of corticosteroids and those of other immunosuppressant medications.

Infliximab will be administered at 5 mg/Kg body weight at 0, 2 and 6 weeks and thereafter, every 2 months for the follow up period of 1 year. Adalimumab will be administered at a dose of 160mg at week 0, 80mg at week 2, 40mg at week 4 and 40mg every other week thereafter.

The outcome of anti-TNF therapy will be evaluated every 2 months and finally at 12 months after the start of therapy. At the same time periods the disease activity will be documented as well. For patients that need dose escalation, the type of dose escalation, i.e. increase in dosing frequency (every one month for infliximab - every week for adalimumab) or increase in dosage (10mg/Kg body weight for infliximab - 80mg for adalimumab) will be recorded. The time from anti-TNF initiation till the need for this dose escalation will also be recorded.

The primary goal of this study is to identify predictors, at baseline, for anti-TNF non-response and anti-TNF loss of response, leading to dose escalation in patients with ulcerative colitis or Crohn's disease that will receive infliximab (CD/UC) or adalimumab (CD) for control of their disease. For this reason at the end of the follow up period (12 months), the following variables will be tested by univariate analysis:

Patient characteristics at baseline

* age
* gender
* weight
* height
* age at onset of disease
* duration of disease until the initiation of anti-TNF therapy
* concomitant corticosteroid use at start of anti_TNF therapy
* concomitant immunosuppresant use at start of anti-TNF therapy
* Blood hemoglobin
* Hematocrit
* White blood cells
* Serum albumin
* C-reactive protein
* ANA
* Anti-ds DNA
* Fecal calprotectin level
* CDAI at baseline for CD patients
* Lichtiger score at baseline for UC patients
* Previous major abdominal surgery
* Tobacco use
* Indication for anti-TNF therapy in CD patients (luminal CD, luminal and fistulizing CD, luminal CD with extraintestinal manifestations)
* Location of disease for CD patients (ileitis, colitis, ileocolitis)
* Location of disease for UC patients (Montreal classification)
* Prior appendectomy
* Family history of IBD

In addition, immunological markers with predictive value for anti-TNF non-response or loss of response will be sought both at intestinal and systemic level. For the determination of mucosal markers, 2 biopsy samples in RNAlater will be collected during the endoscopy prior to the initiation of anti-TNF therapy. Samples will be stored at -80oC and used for the quantitative mRNA expression of various immunological markers, mainly cytokines and their receptors, adhesion molecules and other inflammatory proteins by real time PCR. A third biopsy specimen will be immersed in formalin and maintained for protein expression studies by immunohistochemistry. For the determination of systemic markers, blood will be collected from patients and serum will be separated and stored at -80oC. These samples will be used for the measurement of soluble inflammatory markers that may demonstrate predictive value for anti-TNF non-response or loss of response. Inflammatory markers will be measured by Multiplex assays or by individual ELISAs

ELIGIBILITY:
Inclusion Criteria:

* Active Crohn's luminal ileitis, colitis or ileocolitis necessitating therapy with anti-TNF, according to the physician's judgment, based on the current ECCO guidelines.
* Corticosteroid resistant or corticosteroid dependent ulcerative colitis, necessitating therapy with anti-TNF, according to the physician's judgment, based on the current ECCO guidelines.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: IBD patients treated with anti-TNF that need dose escalation.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Viazis, Principal Investigator — Evangelismos Hospital
Locations (1):
- Evangelismos Hospital, Athens, Greece